CLINICAL TRIAL: NCT00725712
Title: A Phase 2 Study of GSK1363089 (XL880) Administered Orally to Subjects With Metastatic Gastric Cancer
Brief Title: Study of GSK1363089 in Metastatic Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MET111643; NCT00415480 (obsolete NCT alias)
Record Dates: First submitted 2008-07-29; First posted 2008-07-30 (Estimated); Results first posted 2017-08-24 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2016-10

CONDITIONS: Neoplasms, Gastrointestinal Tract
Keywords: c-Met; Metastatic Gastric Carcinoma; adenocarcinoma; Gastric cancer; GSK1363089; XL880; MET inhibitor
MeSH Terms: conditions — Neoplasms; Stomach Neoplasms; Adenocarcinoma | interventions — GSK 1363089

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5-days on/9-days off (Experimental): Dosing for first 5 days in every 14-day period.
  Interventions: Drug: GSK1363089 (formerly XL880)
- daily dosing (Experimental): dosed every day
  Interventions: Drug: GSK1363089 (formerly XL880)

INTERVENTIONS:
Drug: GSK1363089 (formerly XL880) — c-MET tyrosine kinase inhibitor
  Other Names: foretinib

SUMMARY:
This clinical study is being conducted at multiple sites to determine the best confirmed response rate, safety, and tolerability of GSK1363089 treatment in metastatic gastric carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed diagnosis of advanced or metastatic gastric carcinoma, or adenocarcinoma of the gastroesophageal junction or of the distal esophagus. Subjects with tumors of the gastroesophageal junction or of the distal esophagus may be eligible provided that the tumor is not of squamous or sarcomatous histology
* Measurable disease
* The subject consents to provide paired tumor biopsies, directly prior to commencing study treatment and then between Days 5 and 8.
* The subject has an ECOG performance status ≤2.
* The subject is able to ingest the GSK1363089 capsules.
* In the adrenocorticotropic hormone (ACTH) stimulation test, the subject has a serum cortisol level ≥20 μg/dL (552 nmol/L) 30-90 minutes after injection of ACTH.
* The subject has liver, kidney and marrow function.
* The subject is capable of understanding and complying with the protocol and has signed the informed consent document.
* Sexually active subjects (male and female) must use a medically-accepted method of contraception during the course of the study.
* Female subjects of childbearing potential must have a negative serum pregnancy test at screening.
* The subject has had no other diagnosis of malignancy (unless non-melanoma skin cancer or a malignancy diagnosed ≥5 years ago, and has no evidence of disease for 5 years prior to the screening for this study).
* QTc < 470 msec.

Exclusion Criteria:

* The subject has received more than two lines of prior cytotoxic chemotherapy for locally advanced or metastatic disease. For the purpose of this protocol, neoadjuvant therapy would not be considered to be prior cytotoxic chemotherapy. In addition, potential subjects who have received prior treatment with c-MET signaling inhibitor are excluded.
* The subject has received an investigational drug within 14 days of the first dose of study drug.
* The subject has received chemotherapy, immunotherapy, or radiation therapy (to

  ≥25% of his or her bone marrow) within 14 days or has received nitrosoureas or mitomycin C within 6 weeks prior to the scheduled first dose of GSK1363089.
* The subject has AEs due to investigational drugs or other medications administered more than 21 days prior to enrollment that have not recovered to Grade ≤1 using NCI CTCAE v3.0, with the exception of alopecia greater than grade 1.
* The subject has known brain metastases.
* The subject has uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* The subject is pregnant or breastfeeding.
* The subject is known to be positive for the human immunodeficiency virus (HIV).
* The subject has a previously identified allergy or hypersensitivity to components of the GSK1363089 formulation.
* The subject is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2007-03-31; Primary Completion 2009-11-01 (Actual); Study Completion 2009-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (16):
- United States (16):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Stanford, California
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Billings, Montana
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Shah MA, Wainberg ZA, Catenacci DV, Hochster HS, Ford J, Kunz P, Lee FC, Kallender H, Cecchi F, Rabe DC, Keer H, Martin AM, Liu Y, Gagnon R, Bonate P, Liu L, Gilmer T, Bottaro DP. Phase II study evaluating 2 dosing schedules of oral foretinib (GSK1363089), cMET/VEGFR2 inhibitor, in patients with metastatic gastric cancer. PLoS One. 2013;8(3):e54014. doi: 10.1371/journal.pone.0054014. Epub 2013 Mar 14. PMID 23516391
- [Result] Jhawer M, Kindler HL, Wainberg Z, Ford J, Kunz P, Tang L, McCallum S, Kallender H, Shah MA Assessment of two dosing schedules of GSK1363089 (GSK089), a dual MET/VEGFR2 inhibitor, in metastatic gastric cancern (GC): Interim results of a multicenter phase II study J Clin Oncol 2009, 27 (15S), 4502.
- [Result] Jhawer MP, Kindler HL, Wainberg ZA, Hecht JR, Kerr RO, Ford JM, Henderson C, Mueller T, Keer HN, Shah MA Preliminary activity of XL880, a dual MET/VEGFR2 inhibitor, in MET amplified poorly differentiated gastric cancer (PDGC): Interim results of a multicenter phase 2 study. J Clin Oncol, 2008, 26 (15S), Abstr. 4572
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: MET111643 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: MET111643 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: MET111643 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: MET111643 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: MET111643 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: MET111643 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: MET111643 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 74 participants with Metastatic gastric cancer were enrolled in this sequential cohort study at 15 sites in the United States of America. The study was conducted from 23 March 2007 to 20 October 2009.
Groups:
- GSK1363089, Intermittent 5 and 9 Dosing: The eligible participants in this arm were administered GSK1363089 at 240 milligram (mg) per dosing day orally, on 5 days on and 9 days off cycle every 2 weeks for treatment period of 8 weeks. Participants fasted 2 hours before the dose, followed by a glass of water (after the intake of GSK1363089) and continued to fast 1 hour after each dose
- GSK136308, Daily Dosing: The eligible participants in this arm were administered GSK1363089 at 80 mg daily for treatment period of 8 weeks. Participants fasted 2 hours before the dose, followed by a glass of water (after the intake of GSK1363089) and continued to fast 1 hour after each dose. The enrollment in this cohort was started until the enrollment completion in the Intermittent 5 & 9 dosing arm.
Period: Overall Study
Arm/Group | GSK1363089, Intermittent 5 and 9 Dosing | GSK136308, Daily Dosing
Started | 48 | 26
Completed | 0 | 0
Not Completed | 48 | 26
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Progressive disease | 37 | 16
Not completed — Clinical progression not based on RECIST | 0 | 3
Not completed — Adverse Event | 5 | 5
Not completed — Death | 2 | 0
Not completed — Other: Death | 1 | 0
Not completed — Hospitalized, unable to continue | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- GSK1363089, Intermittent 5 and 9 Dosing: The eligible participants in this arm were administered GSK1363089 at 240 mg per dosing day orally( viz. foretinib solid capsules of 20, 100 and 200mg) , as 5 days on and 9 days off cycle (no drug for 9-days) every 2 weeks for treatment period of 8 weeks. Participants fasted 2 hours before the dose, followed by a glass of water (after the intake of GSK1363089) and continued to fast 1 hour after each dose.
- Total: Total of all reporting groups
Arm/Group | GSK1363089, Intermittent 5 and 9 Dosing | GSK136308, Daily Dosing | Total
Number analyzed (Participants) | 48 | 26 | 74
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.1 (12.68) | 59.5 (15.35) | 59.3 (13.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 6 | 19
  Male | 35 | 20 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 42 | 18 | 60
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response Rate (ORR), of GSK1363089, Per- Response Evaluation Criteria in Solid Tumors (RECIST) Criteria Version 1.0
Description: ORR is defined as the percentage of participants achieving best overall response of confirmed complete response (CR) or partial response (PR). Tumor response for participants with measurable lesions was assessed routinely (after 8 weeks of treatment and approximately every 8 weeks thereafter) using RECIST (version 1.0) criteria. The CR for target lesions was defined as disappearance of all target lesions (TLs) and the non-target lesions (NTLs). PR defined as at least 30% decrease in sum of the longest diameter (LD) of TLs, taking as reference baseline sum LD. The safety population included all participants who passed the screening criteria, enrolled in the study, and received at least 1 dose of study drug. Progressive disease will be used as PD.
Time Frame: At every 8 Weeks upto 31 months
Population: Evaluable population included participants from safety population who had received atleast 75% of protocol mandated doses at treatment period, had BL and post BL tumor assessment, with no extended lost to followup (17 wks or more) or who had received atleast 75% of protocol mandated doses at treatment period and discontinued study drug due to PD.
Measure: Number; unit: participants
Arm/Group | GSK1363089, Intermittent 5 and 9 Dosing | GSK136308, Daily Dosing
Number analyzed (Participants) | 44 | 25
participants | 0 | 0

2. Primary Outcome: Number of Participants With Adverse Event (AE) and Serious Adverse Event (SAE)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product whether or not it is considered drug related. This would include any side effect, injury, toxicity, sensitivity reaction, abnormal or worsening of a laboratory value, concurrent illness or sudden death. Pre-existing conditions that worsen during a study will be reported as AEs. SAE is an AE that results in death, is life-threatening, requires inpatient hospitalization or extends a current hospital stay, results in an ongoing or significant incapacity or interferes substantially with normal life functions, or causes a congenital anomaly or birth defect. Medical events that do not result in death, are not life-threatening, or do not require hospitalization may be considered SAEs if they put the participant in danger or require medical or surgical intervention to prevent one of the results listed above.
Time Frame: Up to 31 months
Population: Safety population included all participants who passed the screening criteria, enrolled in the study, and received at least 1 dose of study drug.
Measure: Number; unit: participants
Groups:
- GSK1363089, Intermittent 5 and 9 Dosing: The eligible participants in this arm were administered GSK1363089 at 240 mg per dosing day orally( viz. foretinib solid capsules of 20, 100 and 200 mg) , as 5 days on and 9 days off cycle (no drug for 9-days) every 2 weeks for treatment period of 8 weeks. Participants fasted 2 hours before the dose, followed by a glass of water (after the intake of GSK1363089) and continued to fast 1 hour after each dose.
Arm/Group | GSK1363089, Intermittent 5 and 9 Dosing | GSK136308, Daily Dosing
Number analyzed (Participants) | 48 | 26
participants
  Any AE | 48 | 26
  Any SAE | 22 | 16

3. Primary Outcome: Change From Baseline in Vital Signs-Systolic and Diastolic Blood Pressure
Description: Participants systolic blood pressure (SBP) and diastolic blood pressure (DBP) were measured in mm of mercury (mmHg). These were collected after the participant sat quietly for at least five minutes. The change from baseline was calculated by subtracting the baseline values from the individual post-randomization values. The data for minimum (min) and maximum (max) post-baseline has been reported. Baseline is defined as the last non-missing record on or before first dose.
Time Frame: Baseline (pre-dose, Day 1) and before 30-day follow- up (up to 2 years)
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | GSK1363089, Intermittent 5 and 9 Dosing | GSK136308, Daily Dosing
Number analyzed (Participants) | 48 | 26
mmHg
  SBP, max.post baseline: number analyzed (Participants) | 48 | 25
  SBP, max.post baseline | 25.7 (17.15) | 23.0 (18.87)
  SBP, min.post baseline: number analyzed (Participants) | 48 | 25
  SBP, min.post baseline | -6.3 (18.41) | -5.9 (18.25)
  DBP, max.post baseline: number analyzed (Participants) | 48 | 25
  DBP, max.post baseline | 16.8 (9.21) | 15.4 (9.53)
  DBP, min.post baseline: number analyzed (Participants) | 48 | 25
  DBP, min.post baseline | -3.7 (9.99) | -3.0 (9.65)

4. Primary Outcome: Change From Baseline in Vital Signs-Pulse Rate
Description: The pulse rate or heart rate (HR) for the participant's, were collected after the participant sat quietly for at least five minutes. Baseline evaluations were performed within 72 hours before the first dose. If performed within 24 hours of the first dose, baseline evaluations may serve as the pre-dose Day 1 visit evaluations. The change from baseline was calculated by subtracting the baseline values from the individual post-randomization values. Baseline was defined as pre-dose, Day 1. The HR was measured in beats per minute (bpm). The min and max values have been reported.
Time Frame: Baseline (pre-dose, Day 1) and before 30-day follow- up (up to 2 years)
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | GSK1363089, Intermittent 5 and 9 Dosing | GSK136308, Daily Dosing
Number analyzed (Participants) | 48 | 26
beats per minute
  HR, maximum post baseline: number analyzed (Participants) | 48 | 25
  HR, maximum post baseline | 15.4 (17.16) | 10.7 (11.83)
  HR, minimum post baseline: number analyzed (Participants) | 48 | 25
  HR, minimum post baseline | -9.4 (11.00) | -10.8 (13.17)

5. Primary Outcome: Change From Baseline in Temperature
Description: The body temperature for the participants was assessed. These were collected after the participant sat quietly for at least five minutes. The change from baseline was calculated by subtracting the baseline values from the individual post-randomization values. Baseline is defined as the last non-missing record on or before first dose.
Time Frame: Baseline (pre-dose, Day 1) and before 30-day follow- up (up to 2 years)
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: degree celsius
Groups:
- GSK136308, Daily Dosing: The eligible participants in this arm were administered GSK1363089 at 80 mg daily for treatment period of 8 weeks. Participants fasted 2 hours before the dose, followed by a glass of water (after the intake of GSK1363089) and continued to fast 1 hour after each dose. The enrollment in this cohort was started until the enrollment completion in the Intermittent 5 and 9 dosing arm.
Arm/Group | GSK1363089, Intermittent 5 and 9 Dosing | GSK136308, Daily Dosing
Number analyzed (Participants) | 48 | 25
degree celsius
  Temperature, max.post baseline | 0.46 (0.405) | 2.81 (12.300)
  Temperature, min.post baseline | -0.48 (0.626) | -0.56 (0.629)

6. Primary Outcome: Change From Baseline in Respiratory Rate (RR)
Description: The RR for the participant's, were collected after the participant sat quietly for at least five minutes. Baseline evaluations should be performed within 72 hours before the first dose. If performed within 24 hours of the first dose, baseline evaluations may serve as the pre-dose Day 1 visit evaluations. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. Baseline was defined as pre-dose, Day 1 . The RR was measured in breaths per minute. Min and max post-baseline values are reported.
Time Frame: Baseline (pre-dose, Day 1) and before 30-day follow- up (up to 2 years)
Population: Safety population. Only those participants available at the specified time-points were analyzed.
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | GSK1363089, Intermittent 5 and 9 Dosing | GSK136308, Daily Dosing
Number analyzed (Participants) | 48 | 26
breaths per minute
  RR, maximum post baseline: number analyzed (Participants) | 48 | 25
  RR, maximum post baseline | 1.6 (2.44) | 1.9 (1.89)
  RR, minimum post baseline: number analyzed (Participants) | 48 | 25
  RR, minimum post baseline | -1.3 (1.86) | -1.3 (2.13)

7. Primary Outcome: Number of Participants With Shift From Baseline in by High/Low Flag for Serum Chemistry- Ungraded
Description: The data for serum chemistry parameters like albumin, alanine aminotransferase (ALT), alkaline phosphatase (ALP), amylase, aspartate amino transferase (AST), calcium, carbon dioxide, creatinine, gamma glutamyl transferase (GGT), glucose, blood urea nitrogen (BUN), chloride, free thyroxine, free triiodothyronine, lipase, phosphorous, potassium, sodium, total bilirubin, lactate dehydrogenase, total protein. The abnormal values have been reported wherein data for normal to low and normal to high has been reported.
Time Frame: From Day 1 and before 30-day follow- up (up to 2 years)
Population: Safety population. Only those participants available at the specified time points we re analyzed.
Measure: Number; unit: participants
Arm/Group | GSK1363089, Intermittent 5 and 9 Dosing | GSK136308, Daily Dosing
Number analyzed (Participants) | 48 | 26
participants
  BUN, Normal to low: number analyzed (Participants) | 44 | 24
  BUN, Normal to low | 5 | 1
  BUN, Normal to high: number analyzed (Participants) | 44 | 24
  BUN, Normal to high | 8 | 9
  Chloride, Normal to low: number analyzed (Participants) | 44 | 24
  Chloride, Normal to low | 10 | 3
  Chloride, Normal to high: number analyzed (Participants) | 44 | 24
  Chloride, Normal to high | 5 | 2
  Free Thyroxine , Normal to low: number analyzed (Participants) | 48 | 9
  Free Thyroxine , Normal to low | NA — Data not collected. | 2
  Free Thyroxine , Normal to high: number analyzed (Participants) | 48 | 9
  Free Thyroxine , Normal to high | NA — Data not collected. | 0
  Free Triiodothyronine, Normal to low: number analyzed (Participants) | 48 | 9
  Free Triiodothyronine, Normal to low | NA — Data not collected. | 1
  Free Triiodothyronine, Normal to high: number analyzed (Participants) | 48 | 9
  Free Triiodothyronine, Normal to high | NA — Data not collected. | 0
  Free Triiodothyronine, High to low: number analyzed (Participants) | 48 | 9
  Free Triiodothyronine, High to low | NA — Data not collected. | 1
  Lactate Dehydrogenase, Normal to high: number analyzed (Participants) | 44 | 23
  Lactate Dehydrogenase, Normal to high | 28 | 13
  Protein, Normal to low: number analyzed (Participants) | 44 | 24
  Protein, Normal to low | 7 | 11
  Protein, Normal to high: number analyzed (Participants) | 44 | 24
  Protein, Normal to high | 1 | 0
  TSH, Normal to low: number analyzed (Participants) | 48 | 24
  TSH, Normal to low | NA — Data not applicable. | 0
  TSH, Normal to high: number analyzed (Participants) | 48 | 24
  TSH, Normal to high | NA — Data not applicable. | 7

8. Primary Outcome: Number of Participants With Shift From Baseline in Serum Chemistry- Graded
Description: The worst overall common terminology criteria for adverse events version 3.0 (CTCAE) grade (G) shift post baseline for each parameter was mentioned. Only worst case scenarios are presented. CTCAE grading is done as per intensity namely mild moderate severe life-threatening or Death. Analysis was done for Alanine aminotransferases, aspartate aminotransferases, Albumin, alkaline phosphatase, calcium, sodium, potassium, glucose, amylase, amylase, bilirubin, creatinine, phosphate, gamma glutamyl transferases (GGT), and triglycerol lipase. Worst Overall defined as worst post baseline out of normal range flag in the order of (high, low, normal) before 30 day follow up. Data for G3 and G4 is reported.
Time Frame: From Day 1 to up to 30-day follow-up visit (up to 2 years)
Population: Safety population. Only those participants available at the specified time points were analyzed .
Measure: Count of Participants; unit: Participants
Groups:
- GSK1363089, Intermittent 5 & 9 Dosing: The eligible participants in this arm were administered GSK1363089 at 240 mg per dosing day orally( viz. foretinib solid capsules of 20, 100 and 200mg) , as 5 days on and 9 days off cycle (no drug for 9-days) every 2 weeks for treatment period of 8 weeks. Participants fasted 2 hours before the dose, followed by a glass of water (after the intake of GSK1363089) and continued to fast 1 hour after each dose.
Arm/Group | GSK1363089, Intermittent 5 & 9 Dosing | GSK136308, Daily Dosing
Number analyzed (Participants) | 48 | 26
Participants
  Alanine aminotransferase, G0 to G3: number analyzed (Participants) | 44 | 24
  Alanine aminotransferase, G0 to G3 | 0 | 1
  Alanine aminotransferase, G0 to G4: number analyzed (Participants) | 44 | 24
  Alanine aminotransferase, G0 to G4 | 1 | 0
  Albumin, G0 to G3: number analyzed (Participants) | 44 | 24
  Albumin, G0 to G3 | 0 | 1
  Albumin, G1 to G3: number analyzed (Participants) | 44 | 24
  Albumin, G1 to G3 | 1 | 0
  Albumin G2 to G3: number analyzed (Participants) | 44 | 24
  Albumin G2 to G3 | 1 | 0
  Alkaline phosphatase, G0 to G3: number analyzed (Participants) | 44 | 24
  Alkaline phosphatase, G0 to G3 | 1 | 0
  Amylase, G0 to G3: number analyzed (Participants) | 41 | 21
  Amylase, G0 to G3 | 1 | 0
  Aspartate aminotransferase, G1 to G3: number analyzed (Participants) | 44 | 24
  Aspartate aminotransferase, G1 to G3 | 4 | 0
  Aspartate aminotransferase, G0 to G4: number analyzed (Participants) | 44 | 24
  Aspartate aminotransferase, G0 to G4 | 1 | 0
  Aspartate aminotransferase, G2 to G3: number analyzed (Participants) | 44 | 24
  Aspartate aminotransferase, G2 to G3 | 2 | 0
  Bilirubin, G0 to G3: number analyzed (Participants) | 44 | 24
  Bilirubin, G0 to G3 | 1 | 0
  Creatinine, G0 to G3: number analyzed (Participants) | 44 | 24
  Creatinine, G0 to G3 | 1 | 0
  GGT, G1 to G3: number analyzed (Participants) | 39 | 23
  GGT, G1 to G3 | 3 | 1
  GGT, G2 to G3: number analyzed (Participants) | 39 | 23
  GGT, G2 to G3 | 2 | 0
  Phosphate, G0 to G3: number analyzed (Participants) | 38 | 22
  Phosphate, G0 to G3 | 1 | 0
  Triacylglycerol Lipase, G0 to G3: number analyzed (Participants) | 42 | 22
  Triacylglycerol Lipase, G0 to G3 | 2 | 1
  Triacylglycerol Lipase, G3 to G4: number analyzed (Participants) | 42 | 22
  Triacylglycerol Lipase, G3 to G4 | 1 | 0
  Sodium, G0 to G3: number analyzed (Participants) | 44 | 24
  Sodium, G0 to G3 | 1 | 0
  Sodium, G1 to G3: number analyzed (Participants) | 44 | 24
  Sodium, G1 to G3 | 0 | 1

9. Primary Outcome: Number of Participants With Shift From Baseline by High/Low Flag for Hematology Paramaters
Description: The hematology parameters worst case overall CTCAE grade shift post Baseline for each parameter was mentioned. CTCAE grading for version 3.0 was used and done as per intensity namely mild moderate severe life-threatening or Death. Participants were analyzed for basophils, eosinophils, erythrocytes, hematocrit, and monocytes were analyzed. Only the abnormal values were reported where normal to high and normal to low changes were reported. Worst Overall was defined as highest post baseline CTCAE grade before 30 day follow up.
Time Frame: From Day 1 and before 30-day follow- up (up to 2 years)
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: participants
Arm/Group | GSK1363089, Intermittent 5 and 9 Dosing | GSK136308, Daily Dosing
Number analyzed (Participants) | 48 | 26
participants
  Basophils, Normal to high: number analyzed (Participants) | 44 | 24
  Basophils, Normal to high | 2 | 0
  Eosinophils, Normal to low | 2 | 1
  Eosinophils, Normal to high | 3 | 2
  Erythrocytes, Normal to low | 1 | 2
  Erythrocytes, Normal to high | 1 | 2
  Erythrocytes, Low to high | 0 | 1
  Hematocrit, Normal to low | 3 | 1
  Hematocrit, Normal to high | 3 | 0
  Monocytes, Normal to low | 5 | 3
  Monocytes, Normal to high | 2 | 1

10. Primary Outcome: Number of Participants With Grade Shift for Urinalysis Parameters
Description: The urinalysis parameters by worst case overall CTCAE grade shift post Baseline for each parameter were mentioned as per the CTCAE grading for version 3.0 and done as per intensity namely mild moderate severe life-threatening or Death. Participants were analyzed for abnormal values for bilirubin, ketones, nitrites, occult blood, pH, protein, specific gravity, and urobilinogen.
Time Frame: From Day 1 and before 30-day follow- up (up to 2 years)
Population: Safety population. Only those participants available at the specified timepoints were reported.
Measure: Number; unit: participants
Arm/Group | GSK1363089, Intermittent 5 and 9 Dosing | GSK136308, Daily Dosing
Number analyzed (Participants) | 48 | 26
participants
  Bilirubin, normal to abnormal: number analyzed (Participants) | 39 | 21
  Bilirubin, normal to abnormal | 8 | 3
  Ketones, normal to abnormal: number analyzed (Participants) | 42 | 23
  Ketones, normal to abnormal | 8 | 11
  Nitrites, normal to abnormal: number analyzed (Participants) | 28 | 23
  Nitrites, normal to abnormal | 1 | 1
  Occult blood, normal to abnormal: number analyzed (Participants) | 42 | 23
  Occult blood, normal to abnormal | 11 | 9
  pH, normal to abnormal: number analyzed (Participants) | 42 | 23
  pH, normal to abnormal | 0 | 1
  Protein, normal to abnormal: number analyzed (Participants) | 41 | 22
  Protein, normal to abnormal | 13 | 7
  Specific gravity, normal to abnormal: number analyzed (Participants) | 42 | 23
  Specific gravity, normal to abnormal | 3 | 5
  Urobilinogen, normal to abnormal: number analyzed (Participants) | 34 | 19
  Urobilinogen, normal to abnormal | 3 | 2

11. Primary Outcome: Number of Participants With Shift From Baseline by Grade for Hematology Parameters
Description: The worst overall grading by CTCAE version 3.0, was used to report the shift from baseline for hematology parameters namely hemoglobin, platelets and lymphocytes. The grades were namely G0, G1, G2, G3 and G4. The data for shifts from G2 to G3 and G0 to G4, mainly the shifts to higher grades G3 and G4 have been reported.
Time Frame: Baseline (pre-dose) and before 30-day follow- up (up to 2 years)
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1363089, Intermittent 5 and 9 Dosing | GSK136308, Daily Dosing
Number analyzed (Participants) | 48 | 26
Participants
  Hemoglobin, G2 to G3: number analyzed (Participants) | 44 | 24
  Hemoglobin, G2 to G3 | 0 | 1
  Lymphocytes, G2 to G3: number analyzed (Participants) | 44 | 24
  Lymphocytes, G2 to G3 | 2 | 1
  Platelet, G0 to G4: number analyzed (Participants) | 44 | 24
  Platelet, G0 to G4 | 0 | 1

12. Primary Outcome: Number of Participants Who Required Concomitant Medications
Description: The number of participants who received concomitant medication during the study were reported. The data has been reported for the participants who have received subsequent chemotherapy, subsequent radiation therapy or other therapy.
Time Frame: Baseline (pre-dose) and before 30-day follow- up (up to 2 years)
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1363089, Intermittent 5 and 9 Dosing | GSK136308, Daily Dosing
Number analyzed (Participants) | 48 | 26
Participants
  Subsequent Chemotherapy | 22 | 10
  Subsequent Radiation therapy | 2 | 1
  Other | 1 | 1

13. Secondary Outcome: Median Progression Free Survival (PFS) of GSK1363089
Description: Duration of PFS in months is defined as (Date of Disease Progression/Death - Date of First Dose + 1)/30.44. For participants who did not reach an event (disease progression or death) at the time of data cut-off, duration of PFS is censored at date of last available tumor assessment that is not 'Unable to Evaluate'. For participants who did not have any post-baseline tumor assessments, PFS was censored at Day 1. For any participants who received subsequent anti-cancer therapy, PFS will be right censored at the date of last adequate tumor assessment on or prior to the date of anti-cancer therapy initiation. For any participants who died or progressed after an extended lost-to-follow-up time (greater than 17 weeks), PFS was censored at the date of last adequate assessment prior to extended lost-to follow-up.
Time Frame: At every 8 Weeks upto 31 months
Population: Safety population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | GSK1363089, Intermittent 5 and 9 Dosing | GSK136308, Daily Dosing
Number analyzed (Participants) | 48 | 26
months | 1.64 [1.61 to 1.81] | 1.77 [1.64 to 1.84]

14. Secondary Outcome: Duration of Stable Disease of GSK1363089
Description: Duration of stable disease, was defined as the time between the date of first dose and death or disease progression, in participants whose best overall response was not progressive disease
Time Frame: At every 8 Weeks upto 31 months
Population: Evaluable population. Only those participants available at the specified time-points were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | GSK1363089, Intermittent 5 and 9 Dosing | GSK136308, Daily Dosing
Number analyzed (Participants) | 10 | 5
months | 3.27 [2.92 to 6.11] | 2.69 [1.91 to 3.68]

15. Secondary Outcome: Disease Stabilization Rate of GSK 1363089
Description: It is defined as the number of participants achieving best overall response of confirmed CR or PR or stable disease (SD). It was assessed using RECIST criteria 1.0. The CR for target lesions was defined as disappearance of all TLs and the NTLs. PR is at least 30% decrease in sum of the LD of TLs, taking as reference baseline sum LD. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as a reference, the smallest sum LD since the treatment started.
Time Frame: At every 8 Weeks upto 31 months
Population: Safety population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GSK1363089, Intermittent 5 and 9 Dosing | GSK136308, Daily Dosing
Number analyzed (Participants) | 48 | 26
percentage of participants | 20.8 [10.5 to 35] | 19.2 [6.6 to 39.4]

16. Secondary Outcome: Median Duration of Overall Survival (OS)of GSK1363089
Description: Duration of OS is defined as (Date of Death [due to any cause]) minus Date of first dose. For the participants who were alive at the time of data cut-off, duration of overall survival was censored at the date of last contact. The upper value of the full range was censored observation.
Time Frame: At every 8 Weeks upto 31 months
Population: Evaluable population
Measure: Median (Full Range); unit: months
Arm/Group | GSK1363089, Intermittent 5 and 9 Dosing | GSK136308, Daily Dosing
Number analyzed (Participants) | 44 | 25
months | 7.36 [0.66 to 15.61] | 4.34 [0.79 to 9.23]

ADVERSE EVENTS:
Time Frame: Up to 31 months
Description: Safety population was used for analysis
Groups:
- GSK1363089, Intermittent 5 and 9 Dosing: The eligible participants in this arm were administered GSK1363089 at 240 mg per dosing day orally ( viz. foretinib solid capsules of 20, 100 and 200 mg) , as 5 days on and 9 days off cycle (no drug for 9-days) every 2 weeks for treatment period of 8 weeks. Participants fasted 2 hours before the dose, followed by a glass of water (after the intake of GSK1363089) and continued to fast 1 hour after each dose.
Arm/Group | GSK1363089, Intermittent 5 and 9 Dosing | GSK136308, Daily Dosing
All-Cause Mortality (participants affected / at risk) | 1/48 | 0/26
Serious Adverse Events (participants affected / at risk) | 22/48 | 16/26
Other Adverse Events (participants affected / at risk) | 47/48 | 23/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1363089, Intermittent 5 and 9 Dosing (N=48) | GSK136308, Daily Dosing (N=26)
Disseminated intravascular (Blood and lymphatic system disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Photopsia (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Ascites (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Enterocutaneous fistula (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 5
Obstruction gastric (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Upper gastrointestinal (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 4
Death (General disorders) | 1 | 0
Disease progression (General disorders) | 1 | 2
Fatigue (General disorders) | 2 | 1
Pyrexia (General disorders) | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Alanine aminotransferase (Investigations) | 1 | 0
Aspartate aminotransferase (Investigations) | 1 | 0
Blood alkaline phosphatase (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood urea increased (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Electrocardiogram change (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1363089, Intermittent 5 and 9 Dosing (N=48) | GSK136308, Daily Dosing (N=26)
Nausea (Gastrointestinal disorders) | 18 | 9
Abdominal pain (Gastrointestinal disorders) | 17 | 6
Diarrhoea (Gastrointestinal disorders) | 18 | 5
Vomiting (Gastrointestinal disorders) | 11 | 12
Constipation (Gastrointestinal disorders) | 13 | 8
Dysphagia (Gastrointestinal disorders) | 3 | 5
Abdominal distension (Gastrointestinal disorders) | 6 | 1
Dry mouth (Gastrointestinal disorders) | 3 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3
Ascites (Gastrointestinal disorders) | 3 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 3 | 0
Eructation (Gastrointestinal disorders) | 3 | 0
Flatulence (Gastrointestinal disorders) | 1 | 2
Retching (Gastrointestinal disorders) | 3 | 0
Fatigue (General disorders) | 27 | 15
Oedema peripheral (General disorders) | 11 | 3
Pyrexia (General disorders) | 5 | 4
Mucosal inflammation (General disorders) | 4 | 0
Asthenia (General disorders) | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 13 | 7
Dehydration (Metabolism and nutrition disorders) | 7 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 2
Aspartate aminotransferase increased (Investigations) | 15 | 2
Alanine aminotransferase increased (Investigations) | 11 | 2
Blood lactate dehydrogenase increased (Investigations) | 10 | 2
Weight decreased (Investigations) | 7 | 4
Gamma-glutamyltransferase increased (Investigations) | 8 | 2
Blood alkaline phosphatase increased (Investigations) | 8 | 1
Lipase increased (Investigations) | 1 | 2
Blood creatinine increased (Investigations) | 0 | 2
Headache (Nervous system disorders) | 11 | 3
Dizziness (Nervous system disorders) | 4 | 6
Dysgeusia (Nervous system disorders) | 6 | 0
Paraesthesia (Nervous system disorders) | 4 | 2
Hypoaesthesia (Nervous system disorders) | 3 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 10 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Hypertension (Vascular disorders) | 19 | 4
Deep vein thrombosis (Vascular disorders) | 3 | 0
Hypotension (Vascular disorders) | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 2
Depression (Psychiatric disorders) | 2 | 3
Insomnia (Psychiatric disorders) | 2 | 2
Anxiety (Psychiatric disorders) | 3 | 0
Anaemia (Blood and lymphatic system disorders) | 6 | 1
Dysuria (Renal and urinary disorders) | 3 | 1
Proteinuria (Renal and urinary disorders) | 3 | 0
Urinary tract infection (Infections and infestations) | 5 | 1
Hypothyroidism (Endocrine disorders) | 2 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 | 0
Visual impairment (Eye disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.